CLINICAL TRIAL: NCT04384172
Title: Effect of Peripheral Neuromodulation on Vaginal Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: International Society for the Study of Women's Sexual Health (Unknown); The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, Medical School, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00148746
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Female Sexual Dysfunction; Spinal Cord Injuries
Keywords: peripheral neuromodulation; stimulation; vaginal blood flow
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one arm and completed the other arm 1-5 months later.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tibial nerve stimulation then Genital nerve stimulation (Experimental): Participants who began the study with the tibial nerve stimulation and then proceeded to genital nerve stimulation
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Interventions: Device: Transcutaneous electrical nerve stimulation - Tibial Nerve; Device: Transcutaneous electrical nerve stimulation - Genital Nerve
- Genital nerve stimulation then Tibial nerve stimulation (Experimental): Participants who began the study with the genital nerve stimulation and then proceeded to tibial nerve stimulation
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
  Interventions: Device: Transcutaneous electrical nerve stimulation - Tibial Nerve; Device: Transcutaneous electrical nerve stimulation - Genital Nerve

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation - Tibial Nerve — Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
Device: Transcutaneous electrical nerve stimulation - Genital Nerve — Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.

SUMMARY:
The researchers want to see if nerve stimulation interventions cause a change in vaginal blood flow. This intervention was performed in women who have neurogenic (spinal cord injury) or non-neurogenic sexual dysfunction and healthy women.

DETAILED DESCRIPTION:
Two nerve stimulation locations (genital nerve and tibial nerve) were targeted with skin-surface electrical stimulation in separate experimental sessions.

This study was designed as a crossover study, but all participant data was analyzed together due to small enrollment size.

ELIGIBILITY:
Non-dysfunction participants, no spinal cord injury

Inclusion Criteria:

* Adult (over 18 years old) cis-gender female
* Neurologically stable
* Sexually active at least once per month
* Able to consent and communicate effectively with research team

Exclusion Criteria:

* Male
* Pregnancy or planning to become pregnant during study period
* Sexual dysfunction, per short-form Female Sexual Function Index (FSFI) score below 19
* Lubrication difficulties, per short-form FSFI lubrication subdomain score below or equal to 4
* Clinically diagnosed bladder dysfunction, pelvic pain, or other pelvic organ symptoms
* Suspected or diagnosed epilepsy
* Active infection or active pressure sores in the perineal region
* Implanted pacemaker, defibrillator, spinal cord stimulator, or other nerve stimulator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19.

Sexual dysfunction participants, non- spinal cord injury

Inclusion Criteria:

* Adult (over 18 years old) cis-gender female
* Neurologically stable
* Sexually active at least once per month
* Sexual dysfunction, per short-form FSFI score below 19
* Lubrication difficulties, per short-form FSFI lubrication subdomain score below or equal to 3
* Able to understand consent and communicate effectively with research team

Exclusion Criteria:

* Male
* Pregnancy or planning to become pregnant during study period
* Clinically diagnosed bladder dysfunction, pelvic pain, or other pelvic organ symptoms
* Active infection or active pressure sores in the pelvic region
* Implanted pacemaker or defibrillator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19.

Sexual dysfunction participants with spinal cord injury

Inclusion Criteria:

* Adult (over 18 years old) cis-gender women
* Clinically diagnosed spinal cord injury (AIS A-B) at vertebral level within C6-T10 at least six months prior or clinically diagnosed spinal cord injury (AIS C) at vertebral level within C4-T10 at least six months prior
* Nominally sexually active, but at minimum interest in sexual pleasure even if fully self-induced
* Sexual dysfunction, per short-form FSFI score below 19
* Able to understand consent and communicate effectively with research team

Exclusion Criteria:

* Male
* Spinal cord injury at or above C5 level (C1-C5) if AIS A or B, or spinal cord injury at or above C3 level (C1-C3) if AIS C
* Spinal cord injury below T10 vertebral level or reflexes not preserved
* Acute worsening in motor or sensory function in the last month
* Suspected or diagnosed epilepsy
* Pregnancy or planning to become pregnant during study period
* Active infection or active pressure sores in the perineal region
* Implanted pacemaker or defibrillator
* Currently has or tested positive in the last 14 days for COVID-19 or is symptomatic for COVID-19.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender female
Enrollment: 9 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD at this time.

REFERENCES:
- [Background] Zimmerman LL, Gupta P, O'Gara F, Langhals NB, Berger MB, Bruns TM. Transcutaneous Electrical Nerve Stimulation to Improve Female Sexual Dysfunction Symptoms: A Pilot Study. Neuromodulation. 2018 Oct;21(7):707-713. doi: 10.1111/ner.12846. Epub 2018 Sep 3. PMID 30247794

RESULTS

PARTICIPANT FLOW:
Groups:
- Tibial nerve stimulation then Genital nerve stimulation: Participants who began the study with the tibial nerve stimulation and then proceeded to genital nerve stimulation
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Transcutaneous electrical nerve stimulation - Tibial Nerve: Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Transcutaneous electrical nerve stimulation - Genital Nerve: Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
- Genital nerve stimulation then Tibial nerve stimulation: Participants who began the study with the genital nerve stimulation and then proceeded to tibial nerve stimulation
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
  Transcutaneous electrical nerve stimulation - Tibial Nerve: Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
  Transcutaneous electrical nerve stimulation - Genital Nerve: Standard Transcutaneous electrical nerve stimulation (TENS) device (Empi Select 199584, Medi-Stim Inc.)
  Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
Period: Overall Study
Arm/Group | Tibial nerve stimulation then Genital nerve stimulation | Genital nerve stimulation then Tibial nerve stimulation
Started (Participants who completed their first assigned intervention) | 5 | 4
Washout period (Washout period was one to five months, depending on participant and study team availability) | 5 | 4
Completed (Participants who completed their second assigned intervention) | 4 | 1
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tibial Nerve Stimulation Then Genital Nerve Stimulation | Genital Nerve Stimulation Then Tibial Nerve Stimulation | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Vaginal Pulse Amplitude (VPA) [Mean (Standard Deviation); unit: mV] — While this is shown here in the two arms, data from all participants was analyzed together, regardless of arm.
  VPA will be measured by a vaginal plethysmography transducer. A sensor placed in the vagina will measure changes in blood flow. Population: One participant did not yield VPA data for either session. Participants who did not complete a stimulation session did not have a baseline VPA value for the session that they missed.
  mV
    Tibial Nerve stimulation session: number analyzed (Participants) | 4 | 1 | 5
    Tibial Nerve stimulation session | 14.3 (11.3) | 18.1 (0) | 15.0 (10.0)
    Genital nerve stimulation baseline: number analyzed (Participants) | 3 | 4 | 7
    Genital nerve stimulation baseline | 13.4 (8.6) | 41.2 (42.2) | 29.3 (33.7)
Baseline Heart Rate [Mean (Standard Deviation); unit: bpm] — Population: Participants who did not complete study did not have a baseline measure for the stimulation session that they missed.
  bpm
    Tibial nerve stimulation baseline: number analyzed (Participants) | 5 | 1 | 6
    Tibial nerve stimulation baseline | 70.6 (11.8) | 108 (0) | 76.8 (18.5)
    Genital nerve stimulation baseline: number analyzed (Participants) | 4 | 4 | 8
    Genital nerve stimulation baseline | 68.5 (12.7) | 77.5 (10.1) | 73.0 (11.7)
Baseline Mean Arterial Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Participants who did not complete both sessions did not have a baseline value for the stimulation session that they missed.
  mmHg
    Tibial nerve stimulation baseline: number analyzed (Participants) | 5 | 1 | 6
    Tibial nerve stimulation baseline | 82.4 (6.1) | 75 (0) | 81.2 (6.3)
    Genital nerve stimulation baseline: number analyzed (Participants) | 4 | 4 | 8
    Genital nerve stimulation baseline | 80.3 (7.1) | 71.9 (3.7) | 76.1 (6.9)
Baseline Arousal Score [Mean (Standard Deviation); unit: score on a scale] — Subjective arousal was evaluated by participants using a five point Likert scale, where 1 being no arousal and 5 being greatest arousal. Population: Participants who did not complete both sessions did not have a baseline score for the stimulation session that they missed.
  score on a scale
    Tibial nerve stimulation baseline: number analyzed (Participants) | 5 | 1 | 6
    Tibial nerve stimulation baseline | 1.4 (0.9) | 1 (0) | 1.3 (0.8)
    Genital nerve stimulation baseline: number analyzed (Participants) | 4 | 4 | 8
    Genital nerve stimulation baseline | 1.4 (0.8) | 1.4 (0.8) | 1.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Average Vaginal Pulse Amplitude (VPA) During Stimulation From the Average Baseline Value
Description: VPA will be measured by a vaginal plethysmography transducer. A sensor placed in the vagina will measure changes in blood flow.
Time Frame: Test baseline (approximately minute 0) up to Test completion (approximately minute 60)
Population: Data was analyzed for each treatment, regardless of the order in which the participant received it. One participant did not yield VPA data for either session.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Tibial Nerve Stimulation: Participants received tibial nerve stimulation Transcutaneous electrical nerve stimulation (TENS) - Tibial Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.) Electrical stimulation applied to target the tibial nerve on one leg, with electrodes above the malleolus and on the bottom of the foot
- Genital Nerve Stimulation: Participants received genital nerve stimulation Transcutaneous electrical nerve stimulation (TENS) - Genital Nerve: TENS device (Empi Select 199584, Medi-Stim Inc.) Electrical stimulation applied to target the genital nerve, with electrodes on either side of the clitoris.
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 5 | 7
Percent change | 3.3 (14.2) | 3.5 (26.7)

2. Secondary Outcome: Percent Change in Heart Rate After Stimulation From Baseline
Description: A heart rate monitor (e.g. electrocardiogram or pulse oximetry) will be placed on the participant's arm, hand, or chest (as is appropriate per monitor)
Time Frame: Test baseline (approximately minute 0) up to Test completion (approximately minute 60)
Population: Data was analyzed for each treatment, regardless of the order in which the participant received it.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 6 | 8
percent change | -6.7 (7.1) | 6.0 (13.2)

3. Secondary Outcome: Percent Change in Mean Arterial Blood Pressure During Stimulation From Baseline
Description: A blood pressure monitor will be placed on the participant's arm, hand, or chest (as is appropriate per monitor) to monitor off-target autonomic responses.
Time Frame: Test baseline (approximately minute 0) up to Test completion (approximately minute 60)
Population: Data was analyzed for each treatment, regardless of the order in which the participant received it.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 6 | 8
percent change | 2.3 (4.8) | 5.6 (13.4)

4. Secondary Outcome: Change in Subjective Arousal After Stimulation
Description: Subjective arousal will be evaluated by participants using a five point Likert scale, where 1 being no arousal and 5 being greatest arousal. Values are presented as the average change in arousal score after stimulation, from the baseline measures.
Time Frame: Test baseline (approximately minute 0) up to Test completion (approximately minute 60)
Population: Data was analyzed for each treatment, regardless of the order in which the participant received it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
Number analyzed (Participants) | 6 | 8
score on a scale | 0.5 (1.2) | 1.1 (1.0)

ADVERSE EVENTS:
Time Frame: Up to 10 months
Description: Participants were monitored for AEs during treatments and were given contact information for the study team so they could report AEs that happened after the treatments.
Arm/Group | Tibial Nerve Stimulation | Genital Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04384172/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT04384172/ICF_001.pdf